CLINICAL TRIAL: NCT00489294
Title: An Open-Label Study of the Pharmacokinetics and Pharmacodynamics of Syntropin (a Human Growth Hormone) in Growth Hormone-Suppressed Healthy Volunteers
Brief Title: Safety Study of Syntropin (Human Growth Hormone) for the Treatment of Growth Hormone Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phage Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SYN-05-001
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Growth Hormone Deficiency
Keywords: Human growth hormone; idiopathic short stature; short stature
MeSH Terms: conditions — Dwarfism, Pituitary; Dwarfism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Syntropin

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of Syntropin (a human growth hormone) and to determine the serum concentration of IGF-1 after Syntropin injection.

DETAILED DESCRIPTION:
Syntropin will be administered by subcutaneous injection. Eligible patients will receive a subcutaneous injection of octreodite (to suppress endogenous growth hormone secretion) 12 hours before, immediately prior to, and 12 hours after the scheduled injection of growth hormone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 and 45 years (inclusive).
* Written informed consent to participate in the study.
* Body mass index between 19 and 31 kg/m².
* Female subjects of childbearing potential, defined as not surgically sterile or at least 2 years postmenopausal, must agree to use one of the following forms of contraception from 3 months prior through 7 days following the last dose of study drug: hormonal (oral, transdermal, implant, or injection), barrier (condom, diaphragm with spermicide), IUD, or vasectomized partner (6 months minimum). Subjects must have used the same method for at least 3 months prior to starting the study.
* No clinically significant abnormal findings on the physical examination, medical history, electrocardiogram, or clinical laboratory results during screening.
* Screening growth hormone and insulin-like growth factor I (IGF-I) within normal limits.

Exclusion Criteria

* A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Principle Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* A history of allergic or adverse responses to growth hormone, glycerin, or metacresol, or any comparable or similar product.
* Subjects who (for whatever reason) have been on an abnormal diet during the four weeks preceding the study.
* Subjects who donated blood within 30 days or plasma within 14 days of the first study dosing.
* Participation in a clinical trial within 30 days prior to study initiation.
* Use of any over-the-counter (OTC) medication, including vitamins, within 7 days prior to or during the study.
* Use of any prescription medication within 14 days prior to or during the study, with the exception of hormonal contraceptives for women of childbearing potential.
* Treatment with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to or during the study.
* Smoking or use of tobacco products within 6 months prior to or during the study.
* Female subjects who are trying to conceive, are pregnant, or are lactating.
* Positive serum pregnancy test at screening or urine pregnancy test prior to each drug administration for all women regardless of childbearing potential.
* Positive blood screen for HIV, Hepatitis B surface antigen (HbSAg), or Hepatitis C, or a positive urine screen for alcohol or drugs of abuse.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-08; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics

SECONDARY OUTCOMES:
serum concentrations of insulin-like growth factor-1 (IGF-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States